CLINICAL TRIAL: NCT04950803
Title: A Randomised-controlled Trial of an Oral Microbiome Immunity Formula in Reducing Development of Long-term Co-morbidities in Recovered COVID-19 Patients
Brief Title: A Randomised-controlled Trial of an Oral Microbiome Immunity Formula in Recovered COVID-19 Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RECOVERY
Record Dates: First submitted 2021-06-21; First posted 2021-07-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Probiotic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Subjects will take microbiome immunity formula (SIM01) daily for 6 months
  Interventions: Dietary Supplement: Microbiome immunity formula
- Placebo arm (Placebo Comparator): Subjects will take active vitamin daily for 6 months
  Interventions: Dietary Supplement: Active placebo

INTERVENTIONS:
Dietary Supplement: Microbiome immunity formula — Microbiome immunity formula contains probiotics blend (3Bifidobacteria, 20 billion CFU daily)
  Arms: Active arm
Dietary Supplement: Active placebo — Active placebo contains active vitamin
  Arms: Placebo arm

SUMMARY:
This study aims to evaluate the effectiveness of an oral microbiome immunity formula in modulating gut microbiota, enhancing immunity and reducing long-term complications and co-morbidities in patients who have recovered from COVID-19.

DETAILED DESCRIPTION:
SARS-CoV-2, the cause of COVID-19, emerged as a new zoonotic pathogen of humans at the end of 2019 and rapidly developed into a global pandemic. It may develop severe or critical disease with respiratory failure requiring oxygen support and intensive care.

Natural infection by virus triggers an effective system immunity so that the host can resist or highly reduce the chance of re-infection.

In many cases, this protection can maintain a long period of time. However, the long-term immunities (over a year) and complications from the patients are not yet very clear. We found that COVID-19 survivors who have cleared the virus continued to have persistent altered gut microbiota and up to 80 percent had residue COVID-19 related symptoms including fatigue, difficulty in breathing, impaired memory and hair loss up to 6 months after discharge (LONG COVID-19).

Earlier studies from our CU Medicine have shown a link between altered gut microbiome and COVID-19 severity, and more patients who received a novel microbiome immunity formula (SIM01) achieved complete symptom resolution and developed neutralising antibody than those who did not (unpublished data). Research from the Faculty also reported that almost 40% of people in Hong Kong had significant gut dysbiosis especially in elderly and patients with diabetes, obesity or chronic diseases.

This study is a single-centre, triple-blind, randomized, placebo-controlled clinical trial that aims to evaluate the effectiveness of an oral microbiome immunity formula (SIM01) invented by the Chinese University of Hong Kong (CUHK) in modulating gut microbiota, enhancing immunity and reducing long-term complications and co-morbidities (e.g. sepsis, cardiopulmonary complications, metabolic syndrome, neuropsychiatric disorders) in patients who have recovered from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 and above;
2. Subjects who are mentally capable to participate in the study and provide informed consent;
3. Subjects who can communicate in Chinese or English;
4. Subjects who are ambulatory and do not have difficulties travelling to the clinics for follow-up;
5. Subjects who do not have plans to leave Hong Kong in the subsequent two years after recruitment; and
6. Subjects who agree to give informed consent voluntarily.

Exclusion Criteria:

1. Subjects who are unable to receive oral fluids;
2. Subjects who have received surgery involving the intestine within past 30 days;
3. Subjects who are pregnant or breastfeeding; and
4. Subjects who are immunocompromised, e.g. on cancer treatment, bone marrow/organ transplant, immune deficiency, poorly controlled HIV/AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Alleviation of symptoms or complications | 6 months
  Proportion of subjects with alleviation of symptoms or complication of post-COVID conditions within 6 months.

SECONDARY OUTCOMES:
Any comorbidities | 24 months
  A composite outcome of any comorbidities, including clinical manifestations of long-COVID, hospitalizations due to sepsis, cardiopulmonary complications, metabolic syndrome and neuropsychiatric disorders
Increase in metabolic syndrome (MetS) score | 24 months
  a validated index computed from an analysis based on waist circumference, fasting triglycerides, fasting glucose, and systolic blood pressure, calculated in score (1-5), higher levels indicated higher probability of presence of metabolic syndrome
Increase in other system-specific comorbidities | 24 months
  Increase in other system-specific comorbidities involving cardiovascular, gastrointestinal, liver, renal, genitourinary, haematological, and neurological systems
Healthcare service utilization | 24 months
  The frequency of healthcare service (including clinics and Accident and Emergency) that the subject has attended
Self-reported long-COVID-19 symptoms | 24 months
  Subjects will fill in a survey whether they have long-COVID-19 symptoms (e.g. cough, fatigue, etc) and grade the symptoms. The higher the score, the worse the outcome.
Changes in Quality of life | 48 months
  Changes in Quality of life using visual analogue scale, score ranging 0-100. The higher the score, the better the outcome.
Changes in faecal microbial and bacterial metabolites | 48 months
  Shotgun metagenomics and metabolomics sequencing of faecal samples at baseline and each visit will be used to generate serial gut microbial taxonomic and bacterial functional profiles.
Blood immunity profiles | 24 months
  Inflammatory cytokines in plasma samples will be identified and quantified using human inflammation panel 1 (13-plex) of LEGENDplex

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, Principal Investigator — CUHK-M&T
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Ngai JC, Ko FW, Ng SS, To KW, Tong M, Hui DS. The long-term impact of severe acute respiratory syndrome on pulmonary function, exercise capacity and health status. Respirology. 2010 Apr;15(3):543-50. doi: 10.1111/j.1440-1843.2010.01720.x. Epub 2010 Mar 19. PMID 20337995
- [Background] Li TS, Gomersall CD, Joynt GM, Chan DP, Leung P, Hui DS. Long-term outcome of acute respiratory distress syndrome caused by severe acute respiratory syndrome (SARS): an observational study. Crit Care Resusc. 2006 Dec;8(4):302-8. PMID 17227266
- [Background] Martin JE, Louder MK, Holman LA, Gordon IJ, Enama ME, Larkin BD, Andrews CA, Vogel L, Koup RA, Roederer M, Bailer RT, Gomez PL, Nason M, Mascola JR, Nabel GJ, Graham BS; VRC 301 Study Team. A SARS DNA vaccine induces neutralizing antibody and cellular immune responses in healthy adults in a Phase I clinical trial. Vaccine. 2008 Nov 25;26(50):6338-43. doi: 10.1016/j.vaccine.2008.09.026. Epub 2008 Sep 26. PMID 18824060
- [Background] Modjarrad K, Roberts CC, Mills KT, Castellano AR, Paolino K, Muthumani K, Reuschel EL, Robb ML, Racine T, Oh MD, Lamarre C, Zaidi FI, Boyer J, Kudchodkar SB, Jeong M, Darden JM, Park YK, Scott PT, Remigio C, Parikh AP, Wise MC, Patel A, Duperret EK, Kim KY, Choi H, White S, Bagarazzi M, May JM, Kane D, Lee H, Kobinger G, Michael NL, Weiner DB, Thomas SJ, Maslow JN. Safety and immunogenicity of an anti-Middle East respiratory syndrome coronavirus DNA vaccine: a phase 1, open-label, single-arm, dose-escalation trial. Lancet Infect Dis. 2019 Sep;19(9):1013-1022. doi: 10.1016/S1473-3099(19)30266-X. Epub 2019 Jul 24. PMID 31351922
- [Background] Perera RA, Mok CK, Tsang OT, Lv H, Ko RL, Wu NC, Yuan M, Leung WS, Chan JM, Chik TS, Choi CY, Leung K, Chan KH, Chan KC, Li KC, Wu JT, Wilson IA, Monto AS, Poon LL, Peiris M. Serological assays for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), March 2020. Euro Surveill. 2020 Apr;25(16):2000421. doi: 10.2807/1560-7917.ES.2020.25.16.2000421. PMID 32347204
- [Background] Bonifacius A, Tischer-Zimmermann S, Dragon AC, Gussarow D, Vogel A, Krettek U, Godecke N, Yilmaz M, Kraft ARM, Hoeper MM, Pink I, Schmidt JJ, Li Y, Welte T, Maecker-Kolhoff B, Martens J, Berger MM, Lobenwein C, Stankov MV, Cornberg M, David S, Behrens GMN, Witzke O, Blasczyk R, Eiz-Vesper B. COVID-19 immune signatures reveal stable antiviral T cell function despite declining humoral responses. Immunity. 2021 Feb 9;54(2):340-354.e6. doi: 10.1016/j.immuni.2021.01.008. PMID 33567252
- [Background] Rupp J, Dreo B, Gutl K, Fessler J, Moser A, Haditsch B, Schilcher G, Matzkies LM, Steinmetz I, Greinix H, Stradner MH. T Cell Phenotyping in Individuals Hospitalized with COVID-19. J Immunol. 2021 Apr 1;206(7):1478-1482. doi: 10.4049/jimmunol.2001034. Epub 2021 Feb 8. PMID 33558375
- [Background] Legros V, Denolly S, Vogrig M, Boson B, Siret E, Rigaill J, Pillet S, Grattard F, Gonzalo S, Verhoeven P, Allatif O, Berthelot P, Pelissier C, Thiery G, Botelho-Nevers E, Millet G, Morel J, Paul S, Walzer T, Cosset FL, Bourlet T, Pozzetto B. A longitudinal study of SARS-CoV-2-infected patients reveals a high correlation between neutralizing antibodies and COVID-19 severity. Cell Mol Immunol. 2021 Feb;18(2):318-327. doi: 10.1038/s41423-020-00588-2. Epub 2021 Jan 6. PMID 33408342
- [Background] Hillier TA, Rousseau A, Lange C, Lepinay P, Cailleau M, Novak M, Calliez E, Ducimetiere P, Balkau B; D.E.S.I.R. Cohort. Practical way to assess metabolic syndrome using a continuous score obtained from principal components analysis. Diabetologia. 2006 Jul;49(7):1528-35. doi: 10.1007/s00125-006-0266-8. Epub 2006 May 16. PMID 16752171
- [Background] DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Stat Med. 1994 Jul 15-30;13(13-14):1341-52; discussion 1353-6. doi: 10.1002/sim.4780131308. PMID 7973215
- [Derived] Lau RI, Su Q, Lau ISF, Ching JYL, Wong MCS, Lau LHS, Tun HM, Mok CKP, Chau SWH, Tse YK, Cheung CP, Li MKT, Yeung GTY, Cheong PK, Chan FKL, Ng SC. A synbiotic preparation (SIM01) for post-acute COVID-19 syndrome in Hong Kong (RECOVERY): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2024 Mar;24(3):256-265. doi: 10.1016/S1473-3099(23)00685-0. Epub 2023 Dec 7. PMID 38071990
- See also: WHO website — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Hong Kong Government website — https://www.coronavirus.gov.hk/eng/index.html
- See also: Quality of Life and Long-term Outcomes After Hospitalization for COVID-19. — https://clinicaltrials.gov/ct2/show/NCT04376658?cond=long+covid+outcome&draw=2&rank=2